CLINICAL TRIAL: NCT03624777
Title: Efficacy of the Stroll Safe Outdoor Fall Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Stroll Safe
Record Dates: First submitted 2018-08-07; First posted 2018-08-10 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Accidental Fall; Injury Prevention; Healthy Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stroll Safe Program (Experimental)
  Interventions: Behavioral: Stroll Safe outdoor fall prevention program
- Outdoor Fall Prevention Brochure (Active Comparator)
  Interventions: Behavioral: Outdoor Fall prevention brochure

INTERVENTIONS:
Behavioral: Outdoor Fall prevention brochure — Participants in the wait list control group will initially receive written information only about preventing outdoor falls
  Arms: Outdoor Fall Prevention Brochure
Behavioral: Stroll Safe outdoor fall prevention program — Participants in the treatment group will attend a once a week 7-week outdoor fall prevention program that includes didactic presentations, group discussions/ problem solving, practice in strategy use, and action planning for safe community mobility.
  Arms: Stroll Safe Program

SUMMARY:
This study examines the effectiveness of the Stroll Safe Outdoor Fall Prevention program, a 7-week group based educational intervention. Half of participants are assigned to the Stroll Safe program and half are assigned to a wait list control group that initially receives written information only on outdoor falls prevention.

ELIGIBILITY:
Inclusion Criteria:

Community-dwelling adults age 60 years or older, English speaking, cognitively competent (i.e. have a Montreal Cognitive Impairment score (MOCA) >24), and able to walk outdoors independently with or without a mobility device. In addition, they must answer "yes" to one or more of the following questions: Have you fallen outdoors and hurt yourself in the past year?, Have you fallen outdoors 2 or more times in the past year?, Are you afraid that you might fall outdoors?, Have you had 2 or more stumbles, trips, or slips outdoors in the past month?

Exclusion Criteria:

Less than 60 years of age, living in an institutional setting (e.g. nursing home), non-English speaker, Montreal Cognitive Assessment Score <24, requiring the assistance of another person to walk outdoors, non-ambulatory, an acute health condition that would interfere with participation(e.g. recent fracture, uncontrolled/poorly managed mental health condition, respiratory disease requiring supplemental oxygen), they reply "no" to all of the following questions: Have you fallen outdoors and hurt yourself in the past year?, Have you fallen outdoors 2 or more times in the past year?, Are you afraid that you might fall outdoors?, Have you had 2 or more stumbles, trips, or slips outdoors in the past month?

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2022-05-18 (Actual)

PRIMARY OUTCOMES:
Change in Outdoor Falls Questionnaire (Subscale score for strategy use) | Baseline, following 7-week program, 2 months post program completion
  Measures use of outdoor fall prevention strategies. Range 0-36 with a higher score indicating greater use of fall prevention strategies.
Change in Falls Behavioral Scale for the Older Person (24 item version) | Baseline, following 7-week program, 2 months post program completion
  Measures awareness of and practice of behaviors to protect against falling. Mean score is calculated. Range 1-4, with a higher score indicating safest behaviors.

SECONDARY OUTCOMES:
Change in Falls Self-Efficacy Scale-International | Baseline, following 7-week program, 2 months post program completion
  Measures level of concern about falling. Range 16-64, with a higher score indicating a greater level of concern.
Change in fall diary reports | Baseline, every two weeks until 2 months post program completion
  Participants keep track of trips, slips, and falls on a calendar. Range 0-no limit. Higher number indicates more slips, trips and falls during the two week look back period.

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Chippendale, PhD, OTR/L, Principal Investigator — New York University
Locations (3):
- United States (3):
  - 1199 Norc, New York, New York
  - Warbasse Cares NORC, New York, New York
  - Rochdale Village NORC, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chippendale T, Albert SM, Mahmood A. Efficacy of the Stroll Safe Outdoor Fall Prevention Program: A Randomized Controlled Trial. Gerontologist. 2023 Oct 17;63(9):1556-1565. doi: 10.1093/geront/gnac145. PMID 36148513